CLINICAL TRIAL: NCT01195727
Title: Multiple-Dose Study to Evaluate the Pharmacokinetics, Pharmacodynamics, Safety, and Tolerability of Apixaban in Pediatric Subjects With an Indwelling Central Venous Catheter
Brief Title: Multiple-Dose Study Apixaban in Pediatric Subjects With an Indwelling Central Venous Catheter
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CV185-079
Record Dates: First submitted 2010-09-03; First posted 2010-09-06 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Venous Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism | interventions — apixaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 5A - Apixaban (Low Dose) (Experimental): Group 5: 12 years to <18 years;
  0.66 mg/m² Oral solution, Oral, Twice A Day (BID), 10 days
  Interventions: Drug: Apixaban
- Group 5B - Apixaban (High Dose) (Experimental): Group 5: 12 years to <18 years;
  1.32 mg/m² Oral solution, Oral, Twice A Day (BID), 10 days
  Interventions: Drug: Apixaban

INTERVENTIONS:
Drug: Apixaban
  Other Names: BMS-562247

SUMMARY:
CV185-079 is a multiple dose Apixaban Pharmacokinetics/Pharmacodynamics (PK/PD) study in pediatric subjects. The objective of this study is primarily to study the PK/PD of Apixaban in pediatric subjects with a central venous catheter.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with chronic stable disease with any type of functioning CVC in the upper or lower venous system (e.g., jugular, subclavian; femoral vein) that is anticipated to remain in the subject for the treatment portion of the study.
* > 12 to <18 years of age

Exclusion Criteria:

* Current or recent (within 3 months of study drug administration) gastrointestinal disease or gastrointestinal surgery that, in the opinion of the investigator and the BMS Medical Monitor, could impact the absorption of the study drug
* Active bleeding or high risk of bleeding

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2011-07-26 (Actual); Primary Completion 2012-06-14 (Actual); Study Completion 2012-07-16 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic (PK): Model-derived population & individual PK parameters (e.g., CL/F, Vc/F, KA) used to estimate steady state Cmax & AUC(TAU), Cmin & Tmax in each subject. Population PK model will be developed using plasma concentration vs time data | Days 1, 2, Day 5, 6 or 7 and Day 11

SECONDARY OUTCOMES:
Evidence of anti-Factor Xa confirmed by analysis of anti-Factor Xa PD analysis | Days 1, 2, Day 5, 6 or 7

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (13):
- United States (4):
  - Children'S Hospital Of Orange County, Orange, California
  - Saint Peter'S University Hospital, New Brunswick, New Jersey
  - The Toledo Children'S Hospital, Toledo, Ohio
  - Penn State Hershey Children'S Hospital, Hershey, Pennsylvania
- Belgium (2):
  - Local Institution, Brussels
  - Local Institution, Leuven
- Canada (2):
  - Local Institution, Edmonton, Alberta
  - Local Institution, Ottawa, Ontario
- Mexico (4):
  - Local Institution, Guadalajara, Jalisco
  - Local Institution, Mexico City, Mexico City
  - Local Institution, Mexico, D. F., Mexico City
  - Local Institution, Puebla City, Puebla
- Local Institution, Amsterdam, Netherlands

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx
- See also: BMS Clinical Trial Education Resource — http://www.bms.com/studyconnect/pages/home.aspx